# Myopia Treatment Study 2 (MTS2)

A Randomized Placebo-Controlled Trial of Spectacles with Highly Aspherical Lenslets or 0.05% Atropine to Slow Progression of Myopia in Children

**Statistical Analysis Plan** 

15 July 2025

# **Version History**

This SAP was written with reference to protocol version 1.0. If the protocol is subsequently updated, then this SAP will be reviewed to ensure consistency with the new protocol. The SAP will not be revised unless the protocol changes require modification of the analyses.

| Version | Protocol<br>Version | Author | Approver | Effective<br>Date | Study Stage |
|---|---|---|---|---|---|
| 1.0 | 1.0 | Rui Wu | Wesley<br>Beaulieu | 15 Jul 2025 | The first participant has not yet been enrolled. |

| Version | Revision Description |
|---------|----------------------|
| 1.0 | Original Version |

# **Approvals**

| Role | Digital Signature or Handwritten Signature/Date | |
|---|---|---|
| Author (Statistician) | Rui Wu | Digitally signed by Rui Wu DN: cn-Rui Wu ou-North Wing Reason: I am the author of this document Location: Date: 2025-07-15 09:55-04:00 |
| Approver (Senior Statistician) | Wesley Beaulieu I agree to the terms defined by the placement of my signature in this document 2025-07-15 08:46-04:00 | |

# 1. Study Overview

1

- 2 The primary objective of MTS2 is to compare the effectiveness of 0.05% atropine eye drops
- 3 versus placebo and of HAL lenses vs. single vision lenses for slowing myopia progression
- 4 (change in axial length) over a two-year treatment period in children aged 5 to less than 12 years
- 5 with spherical equivalent refractive error (SER) myopia of 0.75 D to 6.00 D and at least 0.75 D
- 6 myopia in both principal meridians of each eye at the time of enrollment. On-treatment follow-
- 7 up visits are at 6, 12, 18, and 24 months (primary). Randomized treatment stops at 24 months,
- 8 and participants return at 30 months to assess for rebound effects. Complete eligibility criteria
- 9 and study procedures are described in the study protocol.
- 10 Participants will be randomized 1:1:1:1 to placebo eye drops + single vision lenses, 0.05%
- 11 atropine eye drops + single vision lenses, HAL lenses + placebo eye drops, or HAL lenses +
- 12 0.05% atropine eye drops. Randomization is stratified by baseline age (5 to <9 years, 9 to <12
- 13 years). Analyses involving the combination group (HAL lenses +0.05% atropine eye drops) are
- 14 considered exploratory. Sample size has been set at 87 per group (261 total); details are in the
- 15 study protocol.

16

23

24

25

29

# 2. Consistency with the Protocol

- 17 The author of this document has confirmed the analyses described here are consistent with the
- 18 version of the protocol indicated on the version history page except for the following:
- 19 • Flat corneal radius, anterior chamber depth, and lens thickness will not be collected and 20 therefore the analyses of these outcomes have been removed.
- 21 • Monocular amplitude of accommodation will be analyzed at 18 and 30 months in 22 addition to 6, 12, and 24 months.
  - The Barnard unconditional exact test will be used to compare binary safety outcomes instead of the Fisher exact test.
- The adaptive false discovery rate procedure will be used to account for multiplicity in 26 exploratory analyses.
- 27 A subsequent protocol amendment will reflect these changes. Should there be any further
- 28 discrepancy between the associated protocol and this SAP, the content of the SAP shall prevail.

# 3. Statistical Hypotheses

- 30 A test of superiority will be used to evaluate two hypotheses for the change in axial length from
- 31 baseline at the 24-month visit (primary outcome):
- 32 • Between spectacles with single vision lenses + nightly placebo eye drops (hereafter
- 33 PLACEBO group) and spectacles with HAL lenses + nightly placebo eye drop (hereafter
- 34 **HAL** group)
- 35 • Between **PLACEBO** group and spectacles with single vision lenses + nightly atropine
- 36 0.05% eye drop (hereafter **ATROPINE** group)

- 37 Since two treatments with different mechanisms of action are being compared to a shared control
- group, no adjustment for multiplicity is necessary (Section 16).

#### 39 3.1. ATROPINE Versus PLACEBO

- The 0.05% atropine versus placebo eyedrops hypothesis is evaluated in the cohort using single-
- 41 vision lenses.
- Null Hypothesis (H<sub>0</sub>): There is *no difference* in the primary outcome between the PLACEBO group and the ATROPINE group.
- Alternative Hypothesis (H<sub>a</sub>): There *is a nonzero difference* in the primary outcome between the PLACEBO group and the ATROPINE group.

#### 46 3.2. HAL Versus PLACEBO

- 47 The HAL vs. single vision lenses hypothesis is evaluated in the cohort using placebo eye drops.
- Null Hypothesis (H<sub>0</sub>): There is *no difference* in the primary outcome between the PLACEBO group and the HAL group.
- Alternative Hypothesis (H<sub>a</sub>): There *is a nonzero difference* in the primary outcome between the PLACEBO group and the HAL group.

#### 52 4. Outcome Measures

54

56

59

60

68

#### 53 4.1. Primary Efficacy Outcome

• Change in axial length from baseline at 24 months

#### 55 4.2. Secondary Efficacy Outcomes

- Change in spherical equivalent refractive error (SER) from baseline at 24 months
- Change in axial length from baseline at 30 months
- Change in SER from baseline at 30 months
  - Change in axial length from baseline at 18 months
  - Change in SER from baseline at 18 months
- Change in axial length from baseline at 12 months
- Change in SER from baseline at 12 months
- Change in axial length from baseline at 6 months
- Change in SER from baseline at 6 months

#### 4.3. Exploratory Outcomes

- Change in monocular amplitude of accommodation from baseline at 6, 12, 18, 24, and 30 months
  - Change in pupil size from baseline at 6, 12, 18, 24, and 30 months

- Change in axial length over 24 months (area under the curve)
- Change in axial length from 12 to 24 months
- Change in axial length from 24 to 30 months
- Change in SER over 24 months (area under the curve)
- Change in SER from 12 to 24 months
  - Change in SER from 24 to 30 months
  - Child and parent Treatment Impact Questionnaire scores at 6 months and 24 months.

#### 5. Analysis Cohorts

74

75

76

77

78

79

80

81

82

90

- Intention-To-Treat (ITT) Analysis Cohort: all randomized participants, irrespective of treatment received, will be analyzed according to treatment assignment.
- Safety Analysis Cohort: participants who receive at least one dose of the randomly assigned study medication (placebo or 0.05% atropine) or wear the randomly assigned spectacles (HAL or SVL) for any amount of time.

The primary analysis will follow the ITT principle. It will include all randomized participants.

The data from the ITT cohort will be analyzed according to the group to which the participants were assigned through randomization, regardless of treatment received.

#### 86 **6. Visit Windows**

87 For primary, secondary, exploratory, and subgroup analyses, visits must be completed within the

specified visit windows for data to be included. The table below defines the visit windows.

# 89 **Table 1. Analysis Windows**

| Visit | Target Day | Target Window | Analysis Window |
|---|---|---|---|
| 6 months | Randomization + 183 days | ± 2 weeks<br>169 to 197 days | ± 3 months<br>91 to 273 days |
| 12 months | Randomization + 365 days | ± 2 weeks<br>335 to 379 days | ± 3 months<br>273 to 454 days |
| 18 months | Randomization + 548 days | ± 2 weeks<br>534 to 562 days | ± 3 months<br>454 to 638 days |
| 24 months | Randomization + 731 days | ± 2 weeks<br>717 to 745 days | ± 3 months<br>638 to 821 days |
| 30 months | Randomization + 913 days | ± 2 weeks<br>899 to 927 days | ± 3 months<br>821 to 1003 |

# 7. Primary Efficacy Outcome

The average of three separate axial length measurements visits will be calculated for each eye at

baseline and all follow-up visits. If fewer than three measurements are available for an eye at a

- timepoint, the mean of available measurements will be used to calculate the mean axial length
- 94 for each eye. The mean of the right and left eyes will be used for analysis. The change in mean
- axial length from baseline to the 24-month visit will be used as the primary outcome.
- The primary analysis will be a treatment group comparison of change in axial length from
- baseline at 24-month visit, using a longitudinal discrete-time mixed effects model using axial
- 98 length at randomization, 6, 12, 18, and 24 months as the dependent variable and adjusting for age
- 99 to account for confounding due to potential imbalances between groups and to increase statistical
- power.<sup>1,2</sup> Denominator degrees of freedom will be estimated using the Kenward-Roger method
- 101 (DDFM=KR2 in SAS/STAT version 15.2).<sup>3</sup> Non-independence due to repeated measures on the
- same participant will be accounted for using an unstructured covariance matrix. The treatment
- group difference (active treatment placebo) for change in mean axial length from baseline to 24
- months, 95% confidence interval, and P value for the null hypothesis of no difference will be
- calculated based on the model estimates at 24 months. Within-group summary statistics (mean
- and standard deviation) will be calculated from observed data.
- The model assumptions for the mixed model will be assessed qualitatively without formal
- statistical testing. The linearity assumption of the continuous baseline covariates (SER and age)
- will be evaluated using scatterplots (dependent variable versus independent variables and
- residuals versus fitted values). If the assumption of linearity is seriously violated, then a
- transformation or median split will be considered. Normality and homoscedasticity will be
- assessed using plots of residuals (QQ plot, histogram, scatterplot of residuals versus fitted
- values). With equal sample sizes in each treatment group, the assumption of equal variance is not
- critical for the treatment group comparison. If assumptions are seriously violated, then
- alternative, robust approaches will be considered (e.g., M-estimation, generalized linear model
- using the t distribution, and/or heteroscedasticity consistent standard errors). Linearity and
- normality are not expected to be violated given prior experience in a recent study.<sup>4</sup>
- There will be no explicit imputation of outcome data for exams not completed or completed
- outside of the analysis window, as the mixed model will produce an unbiased estimate of
- treatment effect via direct maximum likelihood if the missing outcome data are missing at
- random (MAR). Intercurrent events will be handled using the treatment policy strategy in which
- observed data are used regardless of whether the intercurrent event occurs (e.g., death,
- withdrawal. loss to follow-up, cessation of treatment, receipt of non-randomized treatment,
- 124 etc.).<sup>5</sup>

#### 125 7.1. Sensitivity Analysis

- Sensitivity analyses will be performed to assess the robustness of the primary outcome.
- 127 7.1.1. Complete Case Analysis
- 128 A sensitivity analysis will be conducted to compare the mean change in axial length from
- baseline to 24 months between the treatment groups using an analysis of covariance (ANCOVA)
- model, adjusting for age and baseline axial length. This analysis will be limited to participants
- completing the 24-month visit and will not include imputation for missing data.

#### 132 7.1.2. Tipping Point Analysis

- A multiple imputation with a shift parameter that adjusts the imputed values will be performed
- with treatment group, age, and axial length at randomization, 6, 12, 18, and 24 weeks in the
- imputation model. The imputed data will be estimated from observations in the same treatment
- group (i.e., stratified by treatment group)<sup>6</sup>. A shift will be applied to each group and the
- estimated treatment effect will be displayed as a function of the two shifts. The tipping points
- where the significance changes direction (from significant to non-significant or *vice versa*) will
- be reported and clinical judgement will decide if the tipping points are plausible with a clear
- justification.

# **7.1.3. Confounding**

- 142 Imbalances between groups in important covariates are not expected to be of sufficient
- magnitude to produce confounding. The primary analysis described above includes a pre-
- specified list of covariates identified in prior work as associated with the outcome. As a
- sensitivity analysis, any baseline demographic or clinical characteristics observed to be
- imbalanced between treatment groups will be added as covariates to the analyses of the primary
- outcome. The determination of a meaningful baseline imbalance will be based on clinical
- iudgement and not a p-value. All variables obtained on a continuous scale will be entered into
- the model as continuous variables, unless it is determined that a variable does not have a linear
- relationship with the outcome. In such a case, categorization and/or transformation will be
- explored.

# 152 8. Secondary Efficacy Outcomes

- 153 Secondary outcome will use the ITT analysis cohort and test the null hypothesis between
- treatment groups.

#### 8.1. Change in Spherical Equivalent Error from Baseline at 24 Months

- 156 The mean SER of each eye at baseline and all follow-up visits, measured by the masked
- examiner using cycloplegic autorefraction, will be calculated as the average of the three separate
- readings from autorefraction. If fewer than three readings are available, the average of available
- readings will be used. The mean of the right and left eyes will be used for analysis. The other
- aspects of the analysis are the same as outlined in the primary analyses (Section 5).

#### 161 8.2. Change in Axial Length from Baseline at 30 Months

- The same method described for the primary outcome (Section 5) will be used, but data from 6,
- 163 12, 18, 24, and 30 months will be included in the model.

#### 8.3. Change in Spherical Equivalent Refractive Error from Baseline at 30 Months

- The same method as described in Section 8.1 will be used but with data from 6, 12, 18, 24, and
- 166 30 months included in the model.

# 8.4. Changes in Axial Length and Spherical Equivalent Refractive Error at 6, 12, and 18

168 Months

The same methods described in Section 5 and Section 8.1 will be used.

#### 170 **9. Exploratory Outcomes**

- Exploratory outcomes will use the ITT cohort and test the null hypothesis of no difference
- between treatment groups.

#### 9.1. Change in Monocular Amplitude of Accommodation at 6, 12, 18, 24, and 30 Months

- 174 Change in the monocular amplitude of accommodation at 6, 12, and 24 months will be analyzed
- using a discrete-time longitudinal mixed effects model adjusted for age similar to the primary
- outcome (Section 5).

#### 177 9.2. Change in Pupil Size at 6, 12, 18, 24, and 30 Months

- 178 The change in pupil size at 6, 12, and 24 months will be analyzed using a discrete-time
- longitudinal mixed effects model adjusted for age similar to the primary outcome (Section 7).

#### 9.3. Change in Axial Length Over 24 Months (Area Under the Curve)

- The change in axial length over 24 months (area under the curve) will be calculated and
- compared between treatment groups using the same discrete-time longitudinal mixed effects
- model used for the analyses of the primary outcome (Section 5). The area under the curve can be
- interpreted as a weighted average of the change in axial length at each visit with weights
- proportional to the time between visits. AUC will be calculated by linear combination of model
- estimates using the trapezoidal rule and the following formula:

$$AUC = \sum_{i=1}^{n} \left( \frac{X_i + X_{i+1}}{2} \times m \right)$$

- Where  $X_i$  is the axial length measured at the  $i^{th}$  visit, m is the number of months between visits i
- and i+1, and n is the number of outcome visits included in the analysis. In this analysis there are
- n = 5 visits total: 0, 6, 12, 18, and 24 months. For presentation, AUC will be divided by the
- number of months between baseline and the  $n^{th}$  visit (i.e., 24) so that the value shown will have
- units of millimeters rather than millimeter months.

#### 193 9.4. Change in Axial Length from 12 to 24 Months

- The change in axial length from 12 to 24 months will be calculated and compared between
- treatment groups using the same discrete-time longitudinal mixed effects model used for the
- analyses of the primary outcome (Section 7).

| 197 9.5. Change in Axial Length from 24 to 3 | 97 | 9.5. Unange | ın | Axiai | Length | irom | 24 | το | 30 | <b>Wionths</b> |
|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|

- The change in axial length from 24 to 30 months will be calculated and compared between
- treatment groups using the same discrete-time longitudinal mixed effects model used for the
- analyses of the secondary outcome of change axial length from 24 to 30 months (Section 8.2).

#### 201 9.6. Change in Spherical Equivalent Refractive Error Over 24 Months

- The change in SER over 24 months will be analyzed using the same methods as axial length
- 203 (Section 9.3).

#### 204 9.7. Change in Spherical Equivalent Refractive Error from 12 to 24 Months

- The change in SER from 12 to 24 months will be calculated and compared between treatment
- 206 groups using the same discrete-time longitudinal mixed effects model used for the analyses of
- 207 the secondary outcome in SER (Section 8.1).

#### 208 9.8. Change in Spherical Equivalent Refractive Error from 24 to 30 Months

- The change in SER from 24 to 30 months will be calculated and compared between treatment
- 210 groups using the same discrete-time longitudinal mixed effects model used for the analyses of
- 211 the secondary outcome in SER (Section 8.3).

#### 212 9.9. Treatment Impact Questionnaire

- The Treatment Impact Questionnaire (TIQ) will be used as a quantitative measure to evaluate
- opinions regarding the burdens and impact of the randomized treatment at 6 months and 24
- 215 months (as questions for the child the Child TIQ and the parent themselves the Parent TIQ).
- The Child-TIQ and Parent-TIQ will undergo separate factor analysis to determine the number of
- domains for each TIQ. Each domain will be refined through the evaluation of misfitting items
- and will then be Rasch scored.
- 219 The Rasch scores will be compared between the two treatment groups using a t test to generate a
- mean difference and 95% CI. If assumptions of the t test are seriously violated (normality and
- homoscedasticity) then the Wilcoxon Rank-Sum test with Hodges-Lehmann estimator and 95%
- 222 confidence interval will be used.
- Note that because the TIQ is not administered at baseline (because treatment has not been
- started), there will be no adjustment for baseline score in any analysis.

#### 225 **10.Safety Analyses**

- 226 Safety analyses will be performed among participants who receive at least one dose of their
- randomly assigned study medication (placebo or 0.05% atropine) or wear their randomly
- assigned spectacles (HAL or SVL) for any amount of time. Adverse events will be coded and
- 229 tabulated based on the Medical Dictionary of Regulatory Activities (MedDRA) by treatment

- group. The severity, frequency, and relationship to study treatment will also be tabulated. There
- will be no formal statistical comparison of adverse events.
- The number and proportion of participants experiencing the following outcomes at any time post
- 233 randomization will be tabulated for each group and compared using the Barnard Unconditional
- Exact Test; risk differences and 95% CIs will be estimated using the exact Mid-P method of
- 235 Agresti and Min.<sup>7</sup>:
- Loss of  $\geq$  2 logMAR lines of binocular near visual acuity
- Loss of  $\geq$  2 logMAR lines of monocular distance visual acuity
- 238 These analyses will include all randomized participants without regard to visit completion
- because loss to follow-up is expected to be low based on prior experience in a recent RCT.<sup>4</sup>

#### 240 11.Intervention Adherence

- Adherence to study eyedrops (atropine and placebo eyedrop) and spectacles (SVL and HAL
- lenses) based on calendars brought to each follow-up visit will be tabulated in each treatment
- 243 group.

#### 244 12.Protocol Adherence and Retention

- 245 Protocol deviations and visit completion rates (excluding participant deaths) will be tabulated for
- each treatment group.

# 247 **13.Baseline Descriptive Statistics**

- 248 The baseline characteristics will be tabulated according to treatment group. At a minimum, the
- following will be included:
- 250 Age
- 251 Sex
- 252 Race
- Ethnicity
- Iris color
- Number of biological parents with myopia
- Distance visual acuity in habitual refractive correction
- Axial length
- 258 SER

#### 259 **14.Planned Interim Analyses**

- There are no formal planned interim analyses for this study. The Data and Safety Monitoring
- 261 Committee will review safety and efficacy data approximately every 6 months and can
- recommend stopping the trial if deemed necessary.

### 263 15.Subgroup Analyses

- Subgroup analyses, i.e., assessments of effect modification (interaction), will be conducted for
- 265 the primary outcome, change in axial length at 24 months, and the key secondary outcome,
- 266 change in SER at 24 months. These analyses will be considered exploratory. Subgroup analyses
- will be interpreted with caution, particularly if the corresponding overall analysis does not
- demonstrate a significant treatment group difference. The general approach for these analyses
- will be to add an interaction term for the subgroup factor by treatment into the analysis models
- described in Section 7 and Section 8.1. The P value for an interaction effect will be shown only if
- there are a minimum of 10 observations per level and treatment group. Statistical power for
- detecting interactions is expected to be low. Within-subgroup means, standard deviations,
- adjusted treatment differences, and 95% confidence intervals will be calculated for the following
- 274 factors:
- 275 Sex
- Race/Ethnicity
- Iris color
- 278 o Brown vs not brown
- 279 Age
- $\circ$  5 to <9 vs 9 to <12
- Axial Length
- 282 SER
- For continuous factors, the interaction P value will be calculated using the continuous version
- and within-subgroup means, standard deviations, differences, and 95% confidence intervals will
- be calculated based on a median split.

# 286 **16.Multiple Comparison/Multiplicity**

- For the primary outcome of axial length, two tests of superiority will be conducted: ATROPINE
- vs PLACEBO and HAL vs PLACEBO. The tests will be performed independently, and each will
- be conducted with an alpha level of 0.05.
- 290 Although two pairwise comparisons are being evaluated, there will be no formal adjustment to
- 291 the familywise error rate. Because the primary objective of this trial is to compare each of two
- active treatments (atropine eye drops and HAL lenses), which likely have different mechanisms
- of action, with a shared PLACEBO control group (not with one another), a multiplicity
- adjustment is not needed.<sup>8-10</sup> The risk of a false positive finding with this approach is lower than
- 295 if the two hypotheses were evaluated in two studies with different control groups. 8 The same
- logic applies to secondary, exploratory, safety, and subgroup analyses.
- 297 For the secondary outcomes (Section 8), the familywise error rate will be controlled with a
- 298 hierarchical (i.e., fixed sequence) approach. If the null hypothesis for the primary outcome (axial
- length) is rejected (for either HAL vs PLACEBO or ATROPINE vs PLACBO), then the first
- secondary outcome (change in SER at 24 months) will be compared without further adjustment
- 301 to the type 1 error rate. 11 If the primary outcome null hypothesis is not rejected, then the

- comparison of the change in SER at 24 months will be considered exploratory; a 95% confidence
- interval (without adjustment for multiplicity) will be presented, and a p-value will not be
- presented. Subsequent secondary outcomes will be tested in the order listed in Section 2.
- For exploratory outcomes, the adaptive two-stage step-up procedure of Benjamini, Krieger, and
- Yekutieli<sup>12</sup> will be used to control the false discovery rate at 5% by adjusting both the 95%
- 307 confidence intervals and P values for the analysis of multiple outcomes. The categories/families
- for FDR adjustment will be as follows:

309

- Pupil size and accommodation
- SER and axial length
- Treatment Impact Questionnaire

313

325

326

327

- There will be no formal adjustment for safety analyses because type 2 errors (false negatives) are
- of greater concern than type 1 errors (false positives).
- The adaptive two-stage step up procedure<sup>12</sup> will be used to control the false discovery rate at 5%
- 317 to adjust for multiple subgroup analyses. Both interaction P values and within-group 95%
- confidence intervals will be adjusted; interaction P values and within-group 95% CIs will be
- considered separate families of tests. P values for interactions will only be presented if the
- 320 overall analysis indicates a significant effect.

# **17. Missing Data**

- In general, the procedure for handling missing data is outlined in each section. Where not
- otherwise specified, missing data will be excluded, and only complete cases will be analyzed.

### 324 18.Additional Tabulations and Analyses

- A flow chart accounting for all participants for all visits and phone calls will be developed.
- Visit and phone contact completion rates for each follow-up visit will be tabulated.
- Proportion of participants with a change in myopia of ≥ 0.50 D, ≥ 0.75 D, and ≥ 1.0 D from baseline to 12, 24, and 30 months.
- Proportion of participants with a change in axial length ≥ 0.25 mm, ≥ 0.375 mm, and ≥ 0.50 mm from baseline to 12, 24, and 30 months.

# 19. Exploratory Analyses in COMBINED Atropine + HAL Lenses Group

- Exploratory comparisons between the COMBINED group and the ATROPINE, HAL, and
- PLACEBO groups will parallel the analyses conducted for the ATROPINE vs PLACEBO and
- HAL vs PLACEBO comparisons described above. There comparisons will inform design of
- future studies.

```
337 19.1. Analysis of Main Effects
```

- An exploratory analysis of change in axial length from baseline to 24 months (Section 7) will be
- repeated by pooling across cells in the factorial design (i.e., testing main effects) if the estimated
- interaction effect is less than the hypothesized mean difference of 0.17 mm based on the 95%
- 341 confidence interval (e.g., the 95% CI excludes +/- 0.17 mm). The interaction effect will be
- estimated from a longitudinal mixed effects linear model with independent variables for baseline
- age, atropine (yes vs no), HAL (yes vs no), and the interaction of atropine vs HAL. The
- interaction effect will be tested based on the estimated marginal means as follows:

345

```
-0.17 \ mm < \bar{x}_{PLACEBO+SVL} - \bar{x}_{PLACEBO+HAL} - \bar{x}_{ATROPINE+SVL} + \bar{x}_{ATROPINE+HAL} < 0.17 \ mm
```

347

355

- 348 If the interaction effect is less than the hypothesized mean difference and there is a significant
- main effect for either atropine or HAL (P<.05) in the above analysis of change in axial length,
- then a similar exploratory analysis will be conducted for change in SER from baseline to 24
- months (Section 8.1) but without testing for interaction. The study is expected to have greater
- power to detect differences in axial length than SER; additionally, SER and axial length are
- expected to be highly corrected. Therefore, the test for interaction will be more reliable in the
- axial length analysis.

#### **20.Example Analysis Code**

- 356 The code in the following sections is an example of how analyses may be performed in
- 357 SAS/STAT version 15.2 or a comparable statistical package.

```
358
      20.1. Primary Analysis
359
      proc sort data=visitPts;
360
             by PtID month;
361
      run;
362
363
      proc mixed data=visitPts plots=(VCIRYPANEL);
364
             where month IN (0, 6, 12, 18, 24);
365
             class PtID TrtGroup month;
366
             model meanSER = TrtGroup|month ageRand|month / s ddfm=kr2;
367
             repeated month / type=un subject=PtID r rcorr;
368
             slice TrtGroup*month / diff cl sliceby=month plots=none;
369
      run; title;
370
      20.2. Area Under the Curve Analysis
371
      proc sort data=visitPts;
372
             by PtID month;
373
      run;
374
375
      proc mixed data=visitPts plots=(VCIRYPANEL);
376
             where month IN (0, 6, 12, 18, 24);
```

```
377
             class PtID TrtGroup month Gender;
378
             model meanSER = TrtGroup | month ageRand | month / s ddfm=kr2;
379
             repeated month / type=un subject=PtID r rcorr;
380
             lsmeans TrtGroup*month;
381
             lsmestimate TrtGroup*month "24-m AUC Atropine"
382
                   3 6 6 6 3 0 0 0 0 0 / divisor = 24 cl;
383
             lsmestimate TrtGroup*month "24-m AUC Placebo"
384
                   0 0 0 0 0 3 6 6 6 3 / divisor = 24 cl;
385
             lsmestimate TrtGroup*month "24-m AUC Difference (Atropine - Placebo)"
386
                   3 6 6 6 3 -3 -6 -6 -6 -3 / divisor = 24 cl;
387
      run; title;
388
      20.3. Subgroup Analysis
389
      proc sort data=visitPts;
390
             by PtID month;
391
      run;
392
393
      proc mixed data=visitPts plots=(VCIRYPANEL);
394
             where month IN (0, 6, 12, 18, 24);
395
             class PtID TrtGroup month Gender;
396
             model meanSER = TrtGroup|month ageRand|month Gender|TrtGroup|month / s
397
      ddfm=kr2;
398
             repeated month / type=un subject=PtID r rcorr;
399
             slice TrtGroup*month*Gender / diff cl sliceby=month*Gender plots=none;
400
             lsmestimate trtGroup*month*Gender "Difference of Differences (Interaction)"
401
                   000000001-1 00000000-11;
402
      run; title;
```

#### 21.References

403

434

- Weise KK, Repka MX, Zhu Y, et al. Baseline factors associated with myopia progression and
- 405 axial elongation over 30 months in children 5 to 12 years of age. *Optom Vis Sci.* Oct 1 2024;101(10):619-406 626. doi:10.1097/OPX.000000000002187
- 407 2. Food and Drug Administration. Adjusting for covariates in randomized clinical trials for drugs and biological products: guidance for industry. US Department of Health and Human Services; 2023.
- 409 3. Kenward MG, Roger JH. An Improved Approximation to the Precision of Fixed Effects from
- 410 Restricted Maximum Likelihood. Computational Statistics and Data Analysis. 2009;(53):2583-2595.
- 411 4. Repka MX, Weise KK, Chandler DL, et al. Low-dose 0.01% atropine eye drops vs placebo for
- 412 myopia control: A randomized clinical trial. *JAMA Ophthalmol*. Aug 1 2023;141(8):756-765.
- 413 doi:10.1001/jamaophthalmol.2023.2855
- 414 5. Food and Drug Administration. E9(R1) Statistical Principles for Clinical Trials: Addendum:
- 415 Estimands and Sensitivity Analysis in Clinical Trials. 2021.
- 416 6. Sullivan TR, White IR, Salter AB, Ryan P, Lee KJ. Should multiple imputation be the method of
- 417 choice for handling missing data in randomized trials? *Stat Methods Med Res.* Sep 2018;27(9):2610-2626.
- 418 doi:10.1177/0962280216683570
- 419 7. Fagerland MW, Lydersen S, Laake P. Recommended confidence intervals for two independent
- 420 binomial proportions. Stat Methods Med Res. Apr 2015;24(2):224-54. doi:10.1177/0962280211415469
- 421 8. Howard DR, Brown JM, Todd S, Gregory WM. Recommendations on multiple testing
- adjustment in multi-arm trials with a shared control group. Stat Methods Med Res. May 2018;27(5):1513-
- 423 1530. doi:10.1177/0962280216664759
- 424 9. Juszczak E, Altman DG, Hopewell S, Schulz K. Reporting of Multi-Arm Parallel-Group
- 425 Randomized Trials: Extension of the CONSORT 2010 Statement. Jama. Apr 23 2019;321(16):1610-
- 426 1620. doi:10.1001/jama.2019.3087
- 427 10. Parker RA, Weir CJ. Non-adjustment for multiple testing in multi-arm trials of distinct
- 428 treatments: Rationale and justification. *Clin Trials*. Oct 2020;17(5):562-566.
- 429 doi:10.1177/1740774520941419
- 430 11. Dmitrienko A, D'Agostino RB, Sr. Multiplicity Considerations in Clinical Trials. N Engl J Med.
- 431 May 31 2018;378(22):2115-2122. doi:10.1056/NEJMra1709701
- 432 12. Benjamini Y, Krieger AM, Yekutieli D. Adaptive linear step-up procedures that control the false
- 433 discovery rate. *Biometrika*. 2006;93(3):491-507. doi:10.1093/biomet/93.3.491